CLINICAL TRIAL: NCT03275727
Title: Self-care Programs in Oncology: a Guided Internet-delivered Individually-tailored Acceptance and Commitment Therapy (ACT)-Influenced Cognitive Behavioural Intervention to Improve Psychosocial Outcomes in Breast Cancer Survivors
Brief Title: A Guided Internet-delivered Individually-tailored ACT-influenced CBT Intervention to Improve Psychosocial Outcomes in Breast Cancer
Acronym: INNOVBC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Linkoeping University (Other Government)
Collaborators: Universidade Nova de Lisboa (Other)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INNOVBC
Record Dates: First submitted 2017-09-01; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Breast Neoplasm
Keywords: Breast Cancer; Survivors; Internet intervention; Psychosocial intervention; Acceptance and Commitment Therapy (ACT); Randomized controlled trial
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - iACT-BC experimental group (Experimental)
  Interventions: Behavioral: iACT-BC
- B - Waiting list control group (Other)
  Interventions: Behavioral: iACT-BC

INTERVENTIONS:
Behavioral: iACT-BC — A Guided INternet-delivered Individually-tailored ACT-influenced Cognitive Behavioural INtervention to ImprOVe Psychosocial Outcomes in Breast Cancer Survivors

SUMMARY:
Background: Internet-delivered interventions (IDI) can provide remarkable opportunities in addressing breast cancer (BC) survivors' unmet needs, as they present an effective strategy to improve care coordination and provide access to efficacious, cost-efficient and convenient survivorship care. Nevertheless, research focusing on this field and aiming at improving survivors´ psychosocial needs is scarce and its practical implementation is limited.

Objectives: This study aims at studying BC patients´ and healthcare providers' attitudes towards IDI; exploring BC patients´ unmet support needs and; determining the acceptability, feasibility, efficacy and cost-effectiveness of iACT-BC, a guided internet-delivered individually-tailored ACT-influenced cognitive behavioural intervention designed to improve psychosocial outcomes in BC survivors when compared to treatment as usual. The primary outcomes in this research are anxiety and depression. Secondary outcomes include psychological flexibility, fatigue, insomnia, Sexual dysfunction (SD) and Health Related Quality of Life.

Methods: A multimethod research design will be applied and two consecutive studies will be performed. Study 1 will explore participants´ attitudes towards IDI as well as, BC patients' psychosocial unmet needs by adopting an exploratory cross-sectional study design. Study 2 will investigate the effectiveness and cost-effectiveness of iACT-BC in BC survivors, by implementing a two-arm, parallel, open label, multicentre, waiting list randomized controlled trial.

Expected Results: It is anticipated that iACT-BC will show to be an effective and cost-effective program in improving anxiety, depression, psychological flexibility, fatigue, insomnia, SD and HRQoL in BC survivors, as opposing to a waiting list control under treatment as usual. The results of this research will be published in accordance with CONSORT 2010 and CONSORT-EHEALTH guidelines and should be available for publication in February 2020.

DETAILED DESCRIPTION:
Background: Breast Cancer (BC) ranks as the most frequent and lethal cancer among women, in Portugal. However, advances in cancer detection and treatment contributed to a steady and significant increase in survival over the past years, and 5-year age-standardized relative survival is currently estimated to be 83,4%. This increase translates into a high and growing number of BC survivors, with a considerable proportion of these patients experiencing sequelae of treatment and late effects that can occur immediately to several years after primary treatment ends. Anxiety, depression, fear of recurrence, existential related issues, fatigue, pain, physical and cognitive impairment, tailored information needs, and sexual dysfunction have been reported as the most common unmet support care needs experienced by these women. The answer to these unmet support care needs relies, in part, on delivering comprehensive, highly coordinated, patient-centred care. However, operationalizing such care may prove difficult in a context of competing priorities and constrained health and social care budgets. In this context, connected health, particularly internet-delivered interventions, can provide remarkable opportunities in overcoming the aforementioned constraints, as presenting an effective and innovative healthcare delivery model capable of improving care coordination and providing access to efficacious, cost-efficient and convenient survivorship care. Nevertheless, research focusing on this field and aiming at improving survivors´ psychosocial needs is scarce and its practical implementation is limited.

Objectives: The objectives of this investigation are: studying BC patients´ and healthcare providers' attitudes towards internet-delivered interventions; exploring breast cancer patients´ unmet support care needs and; determining the acceptability, feasibility, effectiveness and cost-effectiveness of iACT-BC, a guided internet-delivered individually-tailored Acceptance and Commitment Therapy (ACT)-influenced cognitive behavioural intervention designed to improve psychosocial outcomes in BC survivors when compared to treatment as usual (TAU) in a waiting list control group (WLC). The primary outcomes in this research are anxiety and depression. Secondary outcomes include psychological flexibility, fatigue, insomnia, sexual dysfunction and Health Related Quality of Life (HRQoL).

Hypotheses: We hypothesize that participants in the intervention group will have improved anxiety, depression, psychological flexibility, fatigue, insomnia, sexual dysfunction and HRQoL, when compared to a WLC.

Methods: A multimethod research design will be applied and two consecutive studies will be performed: Study 1 - Population characterization study and Study 2 - Efficacy and cost-effectiveness study. Study 1 will explore participants´ attitudes towards internet-delivered interventions as well as, BC patients' psychosocial unmet support needs by adopting an exploratory cross-sectional study design. Study 2 will investigate the effectiveness and cost-effectiveness of iACT-BC in BC survivors, by implementing a two-arm, parallel, open label, multicentre, pragmatic, waiting list randomized controlled trial. A Pilot study, mirroring the conditions applied in Study 2 should be performed in order to evaluate the feasibility and acceptability of iACT-BC. Results from this Pilot study should be appraised and inform execution of Study 2

Ethical approval: This study will soon be submitted to evaluation by CNPD and local ethic committees. Authorization to run the study is expected to be received until January 2018.

Expected Results: It is anticipated that iACT-BC will show to be an effective and cost-effective program in improving psychosocial outcomes such as anxiety, depression, psychological flexibility, fatigue, insomnia, sexual dysfunction and HRQoL in BC survivors, as opposing to a WLC under TAU. The results of this research will be published in accordance with CONSORT 2010 and CONSORT-EHEALTH guidelines and should be available for publication in February 2020.

Keywords: Breast Cancer; Survivors; Internet intervention; Psychosocial intervention; Acceptance and Commitment Therapy (ACT); Randomized controlled trial protocol.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Age ≥ 18 years;
* Ability to read and write in Portuguese.
* History of histologically or cytologically confirmed breast cancer with no evidence of metastatic disease.
* An interval ≥ 6 month from primary adjuvant treatment completion (surgery, chemotherapy and/or radiotherapy), except for hormonal therapy.
* Clinically significant symptoms of at least one of the following conditions: anxiety, depression, fatigue, insomnia and/or sexual dysfunction.
* Ongoing regular psychoactive medication only accepted if dosage has been stable during the last 3 months.
* Daily access to the Internet by computer and/or smartphone.
* Ability to use a computer and/or smartphone and the internet.
* No participation on any other interventional study or clinical trial.

Exclusion Criteria:

* Age ≤ 18 years;
* Inability to co-operate and give informed consent.
* Breast cancer not histologically or cytologically confirmed.
* History of other malignancy within the last 5 years.
* Metastasized breast cancer.
* Current severe, uncontrolled systemic disease or mental disorder.
* Absence of clinically significant symptoms.
* Parallel ongoing psychological treatment.
* Ongoing regular psychoactive medication if dosage has been changed during the last 3 months.
* No access to the internet.
* Inability to use a computer and/or smartphone and the internet.
* Parallel ongoing participation in other interventional study or clinical trial.
* Assessment by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female BC survivors
Enrollment: 128 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Depression | Change from baseline to post-intervention (10 weeks after enrollment), Follow-ups at 3, 6 and 12 months
  Patient Health Questionnaire (PHQ-9)
Anxiety | Change from baseline to post-intervention (10 weeks after enrollment), Follow-ups at 3, 6 and 12 months
  Generalized Anxiety Disorder Scale (GAD-7)

SECONDARY OUTCOMES:
Psychological flexibility | Change from baseline to post-intervention (10 weeks after enrollment), Follow-ups at 3, 6 and 12 months
  Cancer Acceptance and Action Questionnaire (Cancer AAQ)
Fatigue | Change from baseline to post-intervention (10 weeks after enrollment), Follow-ups at 3, 6 and 12 months
  Brief Fatigue Inventory (BFI)
Insomnia | Change from baseline to post-intervention (10 weeks after enrollment), Follow-ups at 3, 6 and 12 months
  Insomnia Severity Index (ISI)
Sexual dysfunction | Change from baseline to post-intervention (10 weeks after enrollment), Follow-ups at 3, 6 and 12 months
  Female Sexual Function Index (FSFI)
Health related quality of life - generic measure | Change from baseline to post-intervention (10 weeks after enrollment), Follow-ups at 3, 6 and 12 months
  EORTC QLQC30
Health related quality of life - breast cancer specific measure | Change from baseline to post-intervention (10 weeks after enrollment), Follow-ups at 3, 6 and 12 months
  EORTC QLQBR23

OTHER OUTCOMES:
Participants' attitudes towards internet interventions | Change from baseline to post-intervention (10 weeks after enrollment), Follow-ups at 3, 6 and 12 months
  Attitudes towards internet interventions survey (ATTIS)
Breast cancer patients' unmet support needs | Change from baseline to post-intervention (10 weeks after enrollment), Follow-ups at 3, 6 and 12 months
  Supportive Care Needs Survey Questionnaire (SCNS-SF34)
Intervention cost-effectiveness | Change from baseline to post-intervention (10 weeks after enrollment), Follow-ups at 3, 6 and 12 months
  Questionnaire on Medical consumption and Productivity losses associated with Psychiatric Illness (TIC-P)
Intervention cost-utility | Change from baseline to post-intervention (10 weeks after enrollment), Follow-ups at 3, 6 and 12 months
  EuroQol EQ-5D-5L

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mendes-Santos C, Weiderpass E, Santana R, Andersson G. A guided internet-delivered individually-tailored ACT-influenced cognitive behavioural intervention to improve psychosocial outcomes in breast cancer survivors (iNNOVBC): Study protocol. Internet Interv. 2019 Feb 10;17:100236. doi: 10.1016/j.invent.2019.01.004. eCollection 2019 Sep. PMID 30949435